CLINICAL TRIAL: NCT05732792
Title: Survey Evaluating the Prevalence and the Severity of Feelings of Self-doubt in European Anesthesiologists
Status: Completed | Type: Observational
Sponsor: Université Libre de Bruxelles (Other)
Responsible Party: Principal Investigator, Sarah Saxena, Principal Investigator, Université Libre de Bruxelles
Other Study IDs: AnesthesiaCIPS
Record Dates: First submitted 2023-02-08; First posted 2023-02-17 (Actual); Last update posted 2023-07-21 (Actual); Status verified 2023-07

CONDITIONS: Imposter Syndrome; Anesthesia
MeSH Terms: conditions — imposter syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Anesth-CIPS: The survey is endorsed by the European Society of Anaesthesiology and Intensive Care (ESAIC) and will be distributed from February 2023 onwards to its members for a period of 6 months.
  Interventions: Other: CIPS Survey

INTERVENTIONS:
Other: CIPS Survey — The survey is endorsed by the European Society of Anaesthesiology and Intensive Care (ESAIC) and will be distributed from February 2023 onwards to its members for a period of 3 months.
  Each anesthesiologist's participation to the survey will be voluntary and anonymous individual consent will be implied by the person's willingness to complete the survey.
  The survey will also mention this.
  All surveys will be administered via SurveyMonkey. Surveymonkey allows to build "Health Insurance Portability and Accountability Act" (HIPAA) compliant surveys that follow strict rules around the protection of health information.
  Of note, Surveymonkey is also GDPR (General Data Protection Regulation) compliant.
  Data gathered from the questionnaires will be safely stored on the surveymonkey database. The access to the result database is held by a password that only the authors can use to analyze the data yielded at the end of the survey period.

SUMMARY:
Impostor syndrome is a form of erroneous self-assessment that is defined as the inability to believe that one's success is earnt and that positive outcomes are the result of one's skills.

The syndrome has been described and studied in an array of different populations including the healthcare setting and academic faculty members working in a competitive environment. A scoping review of the imposter syndrome in physicians and physicians in training concluded that low self-esteem, gender, and institutional culture are linked to high rates of imposter syndrome. The fact that this syndrome has been linked to higher rates of burnout is more worrisome. Moreover, this specific syndrome might prevent physicians from acting in certain situations.

Even though Impostor syndrome has been described in doctors across a wide range of specialties, it has yet to be specifically investigated within anesthesiology. We hypothesize that imposter syndrome prevalence will be high in this population due to core attributes of the profession itself.

With this study, the prevalence and severity of imposter syndrome in the European anesthesia profession will be investigated by using the Clance Impostor Phenomenon Scale (CIPS) scale, which will be completed by anesthesiologists and anesthesiology residents members of the European Society of Anesthesiology and Intensive Care.

In parallel, key demographics that are linked to increased severity of the imposter syndrome will also be investigated.

DETAILED DESCRIPTION:
Imposter syndrome is a difficult to grasp concept. Clance and Imes have been the first to label "the inability to internalize success and the tendency to attribute success to external causes such as luck, error or knowing the appropriate individuals" as 'imposter syndrome'. This concept stemmed from the qualitative observation of high achieving women in 1978. Imposter syndrome might be triggered by anxiety, perfectionism, and self-doubt.

Since then, the syndrome has been better described and studied in an array of different populations including academic faculty members in a competitive environment and the healthcare setting. A scoping review of the imposter syndrome in physicians and physicians in training concluded that low self-esteem, gender, and institutional culture are linked to high rates of imposter syndrome. A recent survey study from Villock et al. explored the rate of imposter syndrome and burnout among American medical students and recognized that about half of the female students and a quarter of the male students experience imposter syndrome. Studies in surgery residents, with a response rate of 47%, found that more than three quarter were either significantly or severely affected by the imposter syndrome. Surgery residents are more prone to imposter syndrome than trained ones. More worrisome is the link to burnout.

Most of the studies mentioned used the Clance imposter phenomenon scale (CIPS) to explore the prevalence of imposter syndrome in the population of choice. The CIPS have been validated and used since 1995.

No study has yet explored imposter syndrome among anesthesiologists, though imposter syndrome prevalence might be high in this population due to core attributes of the profession itself. These attributes are likely to depend on the environment in which anesthesiologists evolve. However, performance in clinical work and skills, great interpersonal qualities such as communication skills and good relationship with patients and colleagues are required to excel in our profession. Some of these personal skills have yet to be taught to anesthesiology residents, endorsing imposter syndrome symptoms.

The prevalence and severity of the imposter syndrome in the European anesthesia profession will be studied by using the CIPS scale in anesthesiologists and anesthesiology residents. In parallel, key demographics that are linked to increased severity of the imposter syndrome will be investigated.

Aims The primary aim of this study is to define the prevalence and severity of imposter syndrome among anesthesiologists, which has never been evaluated on a large scale.

The secondary aim of the present study is to identify risk factors associated with imposter syndrome (Gender, age, level of experience, working country, ethnicity, academic work, main activity).

ELIGIBILITY:
Inclusion Criteria:

* Anesthesiologists

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The survey is endorsed by the European Society of Anaesthesiology and Intensive Care (ESAIC) and will be distributed from February 2023 onwards to its members for a period of 3 months.
Sampling Method: Probability Sample
Enrollment: 700 (Actual)
Dates: Start 2023-02-11 (Actual); Primary Completion 2023-05-11 (Actual); Study Completion 2023-05-14 (Actual)

PRIMARY OUTCOMES:
CIPS | 3 months
  The primary aim of this study is to define the prevalence and severity of imposter syndrome among anesthesiologists, which has never been evaluated on a large scale. This will be done through CIPS (Clance Imposter Phenomenon Scale) score.
  (CIPS is a previously validated survey consisting of 20 questions on a 5-point Likert scale that investigate feelings about self-assessment of competency, praise, and success. Levels of severity of imposter syndrome have been described previously. Briefly, if the total score is 40 or less, the respondent has few Impostor characteristics; if the score is between 41 and 60, the respondent has moderate IP experiences; a score between 61 and 80 means the respondent frequently has Impostor feelings; a score higher than 80 means the respondent often has intense IP experiences. The higher the score, the more frequently and seriously the Impostor Phenomenon interferes in a person's life.

SECONDARY OUTCOMES:
Risk factors IP-anesthesia | 3 months
  The secondary aim of the present study is to identify risk factors associated with imposter syndrome (Gender, age, level of experience, working country, ethnicity, academic work, main activity).

CONTACTS AND LOCATIONS:
Locations (1):
- AZ Sint-Jan Brugge Oostende AV, Bruges, Belgium

IPD SHARING:
Plan to Share IPD: Undecided